CLINICAL TRIAL: NCT06561295
Title: Impact of Spontaneous Breathing Trial Timing on Outcomes in Mechanically Ventilated Adult Patients
Brief Title: Optimal Timing for Spontaneous Breathing Trials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Jie Li, Professor, Rush University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24081701
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Respiration, Artificial; Weaning
Keywords: Spontaneous breathing trial; Weaning; Mechanical ventilation duration
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early morning timing of spontaneous breathing trial (No Intervention): Early Morning Group: Patients in this group will undergo their SBTs between 4:00 AM and 5:00 AM, following the traditional early morning schedule used in some ICUs.
- Later morning timing of spontaneous breathing trial (Experimental): Later Morning Group: Patients in this group will have their SBTs scheduled between 8:00 AM and 9:00 AM, closer to the time of day shift rounds.
  Interventions: Other: Later Morning Timing of Spontaneous Breathing Trials

INTERVENTIONS:
Other: Later Morning Timing of Spontaneous Breathing Trials — Later Morning Group: Patients in this group will have their SBTs scheduled between 8:00 AM and 9:00 AM, closer to the time of day shift rounds.
  Arms: Later morning timing of spontaneous breathing trial

SUMMARY:
This study aims to explore how the timing of Spontaneous Breathing Trials (SBTs) affects recovery in adult patients who are on mechanical ventilation in the ICU. SBTs are tests used to determine if a patient is ready to breathe on their own without the help of a ventilator. The study will compare two different timing strategies for these trials: one group of patients will have the test early in the morning, while the other group will have it later in the morning. By observing the outcomes, such as how long patients need to stay on the ventilator, the study hopes to find the best time to perform these trials to help patients recover more quickly and safely.

DETAILED DESCRIPTION:
This study seeks to understand how the timing of Spontaneous Breathing Trials (SBTs) impacts the recovery of adult patients who are on mechanical ventilation in the Intensive Care Unit (ICU). Mechanical ventilation is a life-support technique used for patients who are unable to breathe on their own. The Spontaneous Breathing Trial is a key step in assessing whether a patient is ready to breathe independently and can safely have the ventilator removed.

Currently, there is no universal standard for the best time of day to conduct these trials. Some hospitals perform SBTs early in the morning, while others wait until later in the morning when more staff are available. This study will compare two groups of patients: one group will have their SBTs early in the morning, and the other group will have them later.

The primary goal is to determine whether the timing of these trials affects how long patients need mechanical ventilation, how quickly they can be safely extubated (removal of the breathing tube), and overall recovery outcomes, such as ICU stay and hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21 years or older.
* Patients who have been on mechanical ventilation for more than 48 hours.
* Patients who have completed at least one SBT.

Exclusion Criteria:

* Patients intubated at other hospitals.
* Patients intubated for surgical or interventional procedures.
* Patients receiving venovenous extracorporeal membrane oxygenation (VV-ECMO).
* Patients with a tracheostomy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
mechanical ventilation duration | From enrollment to the end of study at 28 days
  The primary outcome of this study is the duration of mechanical ventilation, which refers to the total number of days a patient remains on a mechanical ventilator in the ICU. This measure begins from the moment a patient is initially placed on the ventilator and continues until the patient is successfully extubated (the breathing tube is removed) and can breathe independently without the need for ventilatory support.

SECONDARY OUTCOMES:
Duration Between SBT Success and Extubation | From enrollment to the end of study at 28 days
  This outcome measures the time interval (in hours) between when a patient successfully passes a Spontaneous Breathing Trial (SBT) and when they are extubated. A successful SBT indicates that the patient is likely ready to breathe independently without mechanical support.
ICU and Hospital Mortality | From enrollment to the end of study at 28 days
  This outcome records the percentage of patients who die while in the ICU or during their overall hospital stay.
ICU and Hospital Lengths of Stay | From enrollment to the end of study at 28 days
  This outcome measures the total number of days a patient remains in the ICU and the hospital from admission to discharge.
Reintubation Rates | From enrollment to the end of study at 28 days
  This outcome measures the percentage of patients who require reintubation within 48 hours of being extubated.
Tracheostomy Rates | From enrollment to the end of study at 28 days
  This outcome records how often tracheostomy procedures are performed on patients who are unable to be weaned from mechanical ventilation via SBTs. A tracheostomy is a surgical procedure to create an opening through the neck into the trachea for long-term ventilatory support.

CONTACTS AND LOCATIONS:
Overall Officials: JIE LI, PhD, Principal Investigator — Rush University
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Due to institution rule

REFERENCES:
- [Background] Roberts KJ. 2022 Year in Review: Ventilator Liberation. Respir Care. 2023 Nov 25;68(12):1728-1735. doi: 10.4187/respcare.11114. PMID 37402584
- [Background] Jung B, Vaschetto R, Jaber S. Ten tips to optimize weaning and extubation success in the critically ill. Intensive Care Med. 2020 Dec;46(12):2461-2463. doi: 10.1007/s00134-020-06300-2. Epub 2020 Oct 26. No abstract available. PMID 33104823
- [Background] Ouellette DR, Patel S, Girard TD, Morris PE, Schmidt GA, Truwit JD, Alhazzani W, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Kress JP. Liberation From Mechanical Ventilation in Critically Ill Adults: An Official American College of Chest Physicians/American Thoracic Society Clinical Practice Guideline: Inspiratory Pressure Augmentation During Spontaneous Breathing Trials, Protocols Minimizing Sedation, and Noninvasive Ventilation Immediately After Extubation. Chest. 2017 Jan;151(1):166-180. doi: 10.1016/j.chest.2016.10.036. Epub 2016 Nov 3. PMID 27818331
- [Background] Roberts KJ, Goodfellow LT, Battey-Muse CM, Hoerr CA, Carreon ML, Sorg ME, Glogowski J, Girard TD, MacIntyre NR, Hess DR. AARC Clinical Practice Guideline: Spontaneous Breathing Trials for Liberation From Adult Mechanical Ventilation. Respir Care. 2024 Jun 28;69(7):891-901. doi: 10.4187/respcare.11735. PMID 38443142